CLINICAL TRIAL: NCT04997525
Title: Estradiol and Progesterone Levels in Early Pregnancy After Natural, Estradiol + Progesterone or Gonadotrophin Stimulated Frozen Embryo Transfer Cycle
Brief Title: Estradiol and Progesterone Levels Following Frozen Embryo Transfer
Acronym: ESTRO-FET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Copenhagen University Hospital at Herlev (Other)
Collaborators: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Pernille Fog Svendsen, DMSc, DMSc, Copenhagen University Hospital at Herlev
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020-001218-39
Record Dates: First submitted 2021-06-22; First posted 2021-08-09 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Estradiol; Progesterone; follitropin alfa; Glycoprotein Hormones, alpha Subunit

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Natural cycle (Active Comparator): These women will follow their natural cycle and receive one injection of hCG for stimulation of ovulation before embryo transfer
  Interventions: Drug: Chorionic Gonadotropin, Alpha
- Estradiol and progesterone (Active Comparator): These women will receive daily estradiol and progesterone tablets/capsules before and after embryo transfer. Treatment will continue until gestational age 9+6
  Interventions: Drug: Estradiol Tablets; Drug: Progesterone
- Gonadotropin (Active Comparator): These women will receive daily gonadotropin injection before embryo transfer. Ovulation will be stimulated using hCG injection.
  Interventions: Drug: Follitropin Alfa; Drug: Chorionic Gonadotropin, Alpha

INTERVENTIONS:
Drug: Estradiol Tablets — Combined with progesterone
  Arms: Estradiol and progesterone
Drug: Progesterone — Combined with estradiol
  Arms: Estradiol and progesterone
Drug: Follitropin Alfa — Combined with hCG
  Arms: Gonadotropin
Drug: Chorionic Gonadotropin, Alpha — In either natural cycle or combined with Follitropin Alfa
  Arms: Gonadotropin; Natural cycle

SUMMARY:
The aim of the present study is to investigate serum estradiol and progesterone levels in women conceiving after natural, estradiol + progesterone or gonadotropin stimulated frozen embryo transfer (FET) cycles.

DETAILED DESCRIPTION:
Enrolled women will be randomized based on their ovulation pattern. Ovulatory women will be randomized to either natural cycle or estradiol + progesterone substituted cycle treatment for FET. Anovulatory women will be randomized to either estradiol + progesterone substituted cycle or gonadotropin stimulated cycle treatment for FET.

Included women will undergo blood testing every two weeks for serum estradiol and progesterone levels until gestational age 9+6. Routine vaginal ultrasounds will be performed as well as additional pregnancy ultrasounds.

Secondary obstetric outcomes will be investigated using the womens medical journals.

All the treatments are considered standard treatments for FET.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years < 40 years
* BMI < 35 kg/m2
* Normal wet smear within the past three years
* Thawed blastocysts (day 5 or 6) after either IVF or ICSI treatment

Exclusion Criteria:

* Age < 18 years
* BMI > 35 kg/m2
* Oocyte donation
* HIV/ hepatitis
* Undiagnosed vaginal bleeding
* Uterine malformations
* Persisting ovarian cysts
* Tumors in Hypothalamus, pituitary, thyroid or adrenal
* Previous breast cancer
* BRCA1/2
* Unregulated thyroid disease
* Cardiovascular disease
* Breast feeding
* Present or previous chemotherapy/radiation therapy
* Present or previous malignant disease
* Smoking
* Alcohol/drug abuse

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 305 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Serum estradiol | 10 weeks
  Blood samples in the first 10 weeks of pregnancy
Serum progesterone | 10 weeks
  Blood samples in the first 10 weeks of pregnancy

SECONDARY OUTCOMES:
Gestational age at delivery | At delivery
  Weeks of pregnancy when the child has been delivered
Child birth weight | At delivery
  Weight of the child at delivery
Obstetric complications | 9 months
  Obsteric complication throughout pregnancy
Child malformations | 9 months
  Child malformations diagnosed in utero or at delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev University Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No